CLINICAL TRIAL: NCT01526187
Title: Acquisition of Multidrug-resistant Bacteria After Travel in the Tropics : Prevalence, Determinants and Length of Carriage
Brief Title: Travel in the Tropics and Acquisition of Multidrug-resistant Bacteria (VOYAG-R)
Acronym: VOYAG-R
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 11012 (AOR 11101)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2013-03

CONDITIONS: Fecal Carriage of Multidrug-resistant Bacteria
Keywords: Public Health and Epidemiology; Bacteriology; Infectious and Tropical
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Sub-Saharan Africa
- Asia
- Latin America

SUMMARY:
The purpose of this study is to Measure the fecal carriage of multidrug-resistant bacteria after a travel in the tropics.

DETAILED DESCRIPTION:
Bacterial multidrug resistance has long been a hospital problem. This changed in the last decade with the emergence in the community of Enterobacteriaceae producing CTX-M-type extended spectrum beta-lactamases (ESBL). These enzymes are produced mainly by Escherichia coli, the main digestive commensal bacteria in Man, and the first causative agent of community-acquired infections. These strains were isolated in the world with a very high community prevalence in the countries in the tropics, but still low in industrialized countries such as France. The steady increase in international tourism has created daily flux between these areas that could well be a major vehicle for ESBL. While we just reported in Europe Enterobacteriaceae resistant to almost all antibiotics, including production of NDM-1 carbapenemase, imported from the Indian subcontinent is urgently needed to control this phenomenon, quantify and characterize the acquisition of multidrug-resistant Enterobacteriaceae (MRE) by French travelers in the tropics.

Assumptions Travel in the tropics is a source of import of MRE in France.

Population concerned Adult volunteers in the vaccination center prior to a travel in the tropics.

Main objective Measured independently for each of the three main tropical areas (Latin America, Sub-Saharan Africa and Asia) the rate of acquisition of MRE intestinal (for production of ESBL, and / or cephalosporinase plasmid and / or of carbapenemase) in people returning from a trip to the tropics that led to early consultation in a vaccination center.

Objective (s) school (s)

1. - Comparison of MRE acquisition rate in travelers returning by visited region.
2. - Determine the risk factors for acquisition of the MRE during the stay
3. - Measure the length of the MRE carriage after the return of the trip
4. - To study the dynamics of the concentration of MRE in digestive carriers in the stool
5. - To study the influence of antibiotics on the duration of carriage of the MRE
6. - Estimating the occurrence of infections among patients MRE
7. - To identify the genes responsible for multidrug resistance phenotype in MRE
8. - To assess the phylogenetic relationships of the resistant MRE

Primary endpoint The primary endpoint is defined by the presence of MRE in the stool back from traveling in the tropics in patients who were not carriers before travel.

Keyword (s) of secondary assessment (s)

1. - Location: Asia, Sub-Saharan Africa, Latin America
2. - Acquisition of data: sex, age, socioeconomic status, diet, frequency of history of travel in the same geographical area, type of antimalarial prophylaxis (and compliance), type of stay, occurrence of diarrhea, intake antibiotics, contact a health facility during the stay.
3. - Presence of MRE 1, 2, 3, 6 and 12 months after return.
4. - Amount of MRE per gram of stool in each sample
5. - Antibiotics (name and date taken antibiotics) between sending stool.
6. - Report of urinary tract infections occurring during the MRE inclusion of the subject.
7. - Presence of resistance genes by molecular techniques (PCR, sequencing).
8. - Phylogenetic relationships of MRE (Escherichia coli and Klebsiella pneumoniae) assessed by the method of multi-locus sequence typing (MLST).

Type of study Prospective cohort study, multicenter, observational with a stratified sampling of the geographical area of destination (Asia, Sub-Saharan Africa, Latin America).

Methodology Adults consultant in a vaccination center of one of the six investigator wards, prior to a holiday in the tropics are approached by an investigator to participate in the study. The volunteers will send by mail to the laboratory a stool sample in the weeks prior to departure and another within 72 hours after return from which will be investigated and quantified the MRE. Data will be collected by the investigator and then by a self-administered questionnaire to establish risk factors for acquiring MRE during the stay. If positive, follow-up (1, 2, 3, 6, 12 months) will be undertaken to measure the duration of carriage and the dynamics of the concentration of MRE in the stool after the return. The occurrence of urinary tract infections MRE will be recorded. Subjects will be indemnified according to the number of samples sent.

Number of persons needed To analyze a dozen potential risk factors must be provided about 110 events. With an acquisition rate estimated at 20%, 570 subjects analyzed are needed. The inclusion of 750 subjects, of which 5% will probably be excluded as carriers of MRE before the trip and 20% will be lost sight of, will achieve this goal of 570 subjects analyzed. The inclusion of 250 subjects (190 analyzed) in each of three geographical areas (Asia, Latin America, Sub-Saharan Africa), will estimate the rate of acquisition zone with an accuracy of about 5%.

Inclusion Criteria

* Age greater than 18 years
* Consulting a vaccination center
* Travel in the tropics for a minimum of 2 days and maximum of 90 days

Key non-inclusion criteria

* Pregnant woman (known pregnancy) or breastfeeding
* Refusal to participate in the study,
* Accompanied by a subject already included,
* Subject has already been included in the study,
* Inability to follow in the weeks following the return trip in the tropics.

Study Schedule Phase of implementation: 60 days (September 7 to November 7, 2011)

Inclusion period (February 7, 2012 to February 9, 2013) Follow-up period (March 7, 2012 to May 7, 2014) Period of phenotypic analysis of samples (7 February 2012 to May 7, 2014) Period molecular analysis of samples (7 February 2012 to May 7, 2014) Analysis of results (Winter 2013-2014) Publication of results (second half of 2014)

Number of participating centers: 6

Average number of inclusions per month per center: 11

Tags thesaurus DRCD09-V3 (3 maximum):

Public Health and Epidemiology Bacteriology Infectious and Tropical

An ancillary study aims to make a molecular analysis of intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Consulting a vaccination center
* Travel in the tropics for a minimum of 2 days and maximum of 90 day

Exclusion Criteria:

* Pregnant woman (known pregnancy) or breastfeeding
* Refusal to participate in the study,
* Accompanied by a subject already included,
* Subject has already been included in the study,
* Inability to follow in the weeks following the return trip in the tropics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers in the vaccination center prior to a travel in the tropics.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined by the presence of MRE in the stool back from traveling in the tropics in patients who were not carriers before travel. | 12 months

SECONDARY OUTCOMES:
Location, acquisition of data regarding travel conditions and traveller's profile | 12 months
  1. - Location: Asia, Sub-Saharan Africa, Latin America
  2. - Acquisition of data: sex, age, socioeconomic status, diet, frequency of history of travel in the same geographical area, type of antimalarial prophylaxis (and compliance), type of stay, occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Sophie MATHERON, MD,PHD, Principal Investigator — APHP
Locations (1):
- Hôpital BICHAT - CLAUDE BERNARD, Paris, France

REFERENCES:
- [Derived] Armand-Lefevre L, Rondinaud E, Desvillechabrol D, Mullaert J, Clermont O, Petitjean M, Ruppe E, Cokelaer T, Bouchier C, Tenaillon O, Ma L, Nooroya Y, Matheron S, The Voyag-R Study Group, Andremont A, Denamur E, Kennedy SP. Dynamics of extended-spectrum beta-lactamase-producing Enterobacterales colonization in long-term carriers following travel abroad. Microb Genom. 2021 Jul;7(7):000576. doi: 10.1099/mgen.0.000576. PMID 34279212
- [Derived] Ruppe E, Armand-Lefevre L, Estellat C, Consigny PH, El Mniai A, Boussadia Y, Goujon C, Ralaimazava P, Campa P, Girard PM, Wyplosz B, Vittecoq D, Bouchaud O, Le Loup G, Pialoux G, Perrier M, Wieder I, Moussa N, Esposito-Farese M, Hoffmann I, Coignard B, Lucet JC, Andremont A, Matheron S. High Rate of Acquisition but Short Duration of Carriage of Multidrug-Resistant Enterobacteriaceae After Travel to the Tropics. Clin Infect Dis. 2015 Aug 15;61(4):593-600. doi: 10.1093/cid/civ333. Epub 2015 Apr 22. PMID 25904368